CLINICAL TRIAL: NCT05384990
Title: Neuromotor Control During Postural Transitions in Children and Young Adults With Cerebral Palsy
Brief Title: Sensorimotor Control During Postural Transitions in CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Samuel Lee, Director and Associate Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1759703
Record Dates: First submitted 2022-05-11; First posted 2022-05-23 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
Keywords: Balance Control; Stochastic Resonance; Postural Transitions
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Cross sectional study in children with CP and age matched TD (typical developing). Each group will undergo two stimulation conditions, stochastic resonance (SR) stimulation and a no stochastic resonance (noSR) condition while performing postural Transitions.
Who Masked: Participant
Masking Description: The SR stimulation will be provided to the participant in a randomized order using a computer based program. Participants will be unaware of the test condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stochastic Resonance stimulation (Experimental): During this condition, participants will perform postural transitions like sit to stand, gait initiation, sit to walk and Timed Up and Go test while receiving stochastic resonance stimulation on legs and hip.
  Interventions: Device: Stochastic Resonance Electric Stimulation
- No Stochastic Resonance stimulation (No Intervention): During this condition, participants will perform postural transitions like sit to stand, gait initiation, sit to walk and Timed Up and Go test without receiving any electrical stimulation.

INTERVENTIONS:
Device: Stochastic Resonance Electric Stimulation — Subjects will be asked to perform postural transitions like sit to stand, gait initiation, sit to walk and Timed up and the Go (TUG) functional test. This will entail a subsensory electrical signal with a white noise frequency distribution. Proprioceptive SR electrical stimulation will be delivered by BIOPAC Systems, Inc. stimulators that are current limited to deliver less than 10 milli ampere of current. Electrical stimulation will be delivered to muscles and joints along the legs and hips. The stimulation intensity will be very low, below the sensory threshold of the participant.
  Arms: Stochastic Resonance stimulation

SUMMARY:
The purpose of this study is to investigate whether a light electrical stimulation to leg muscles and joints can help people with Cerebral Palsy (CP) maintain balance during everyday tasks such as getting up from a chair and walking. Children and young adults with CP can have trouble with daily tasks such as standing up, sitting down on the chair and turning. The difficulty in maintaining balance sometimes lead to falls. This raises risk of disability in CP as children age into teens and adults. Current treatments are not very effective. In this study, children and young adults will be asked to stand up from a stool, walk in a straight line, turn, walk back and sit down on the stool. Participants will receive electrical stimulation at a very low intensity that cannot be felt to help increase their sensory perception. The investigators will evaluate treatment by testing balance, and other functional measures.

ELIGIBILITY:
Inclusion Criteria for individuals with CP:

1. Age 10-21
2. Diagnosis of CP
3. GMFCS level I-II
4. Ability to stand up from a chair and start walking.
5. Migration index of proximal hip (MIGR) < 40% femoral head covering in acetabulum
6. At least 0° passive dorsiflexion range of motion (ROM)
7. Sufficient visuoperceptual, cognitive and communication skills
8. Seizure-free or well-controlled seizures
9. No other neurological or musculoskeletal disorders (e.g. dystonia, severe scoliosis, hip instability
10. Ability to communicate pain or discomfort
11. Ability to assent/consent or obtain parent/guardian consent

Exclusion Criteria for individuals with CP:

1. Scoliosis with primary curve > 40%
2. Spinal fusions extending into pelvis
3. Lower Extremity joint instability or dislocation
4. Severe tactile hypersensitivity
5. Lower extremity botulinum injections in the past 6 months
6. Implanted medical device or metal contraindicative of the application of SR
7. Pregnancy (self-reported)
8. Severe lower extremity spasticity (Modified Ashworth Scale score of 4 or greater)
9. History of pulmonary disease limiting exercise tolerance (Asthma Control Test screen)
10. History of cardiac disease (American Heart Association screen)
11. Severely limited range of joint motion/ irreversible muscle contractures
12. Lower extremity surgery or significant injury within last 1 yr.

Inclusionary criteria for typically developing volunteers:

1. Aged 10-21 years old
2. Ability to stand up from a chair and start walking without an assistive device or orthoses
3. Able to communicate discomfort during testing and can follow multi-step directions
4. Has not been diagnosed with any neurological or balance disorders
5. Seizure-free

Exclusionary criteria for typically developing volunteers:

1. Diagnosis of CP
2. Significant scoliosis with primary curve > 40°
3. Lower extremity surgery or fractures in the year prior testing
4. Joint instability or dislocation in the lower extremities
5. Severe tactile hypersensitivity
6. A history of selective dorsal root rhizotomy
7. Botulinum toxin injections in the lower extremities within the past 6 months
8. Marked visual or hearing deficits
9. Any embedded metal that may be contraindicated with application of SR
10. Severe spasticity of the lower extremity muscles (eg. a score of 4 on the Modified Ashworth)
11. Pregnancy (self-reported)
12. Severely limited joint range of motion/ irreversible muscle contractures that would not be candidates for soft-tissue surgery
13. Learning disabilities
14. History of neurological disorders
15. Balance and/or postural impairment

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in COM | 2 assessment points: Baseline - pre stimulation COM, and at the end of the session with stimulation (Day 1)- Post stimulation COM
  Change in the Center of Mass (COM) trajectories while performing various activities.
Change in COP | 2 assessment points: Baseline - pre stimulation COP, and at the end of the session with stimulation (Day 1)- Post stimulation COP
  Change in the Center of Pressure (COP) trajectories while performing various activities.
Total time | Baseline, Post Stimulation (Day 1)
  Time taken to complete the task.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lee, PT, PhD, Principal Investigator — University of Dealware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided